CLINICAL TRIAL: NCT02463916
Title: The ExMET-IBD Study: A Randomized Control Trial to Determine the Effects of Exercise on Intestinal Microbiota and Immunological Markers in Patients With Inflammatory Bowel Disease and Rheumatoid Arthritis
Brief Title: A Trial to Determine the Effects of Exercise in Inflammatory Bowel Disease and Rheumatoid Arthritis
Acronym: ExMET-IBD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Professor Fergus Shanahan, Professor and Chair Department of Medicine and Director Alimentary Pharmabiotic Centre, University College Cork, University College Cork
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: APC056
Record Dates: First submitted 2015-03-10; First posted 2015-06-04 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Inflammatory Bowel Disease; Rheumatoid Arthritis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Arthritis, Rheumatoid | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate exercise (Active Comparator): This group will immediately commence an 8 week exercise programme.
  Interventions: Other: Exercise
- Delayed exercise (Active Comparator): This group will continue regular activities for 8 weeks and then commence 8 week exercise programme.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — 8 week structured exercise programme

SUMMARY:
The purpose of this study is too determine the effects of exercise on the gut microbiota and immunological markers in patients with inflammatory bowel disease and rheumatoid arthritis.

DETAILED DESCRIPTION:
Background:

The benefits of exercise are plentiful (1). They are physical, psychological and social. Exercise exhibits its effects on multiple systems through multiple mechanisms. These mechanisms are often poorly understood. Long-term resistance training results in many health benefits. It is associated with a reduced risk of low-grade inflammatory diseases, improved metabolic profile in patients with type two diabetes and the prevention of osteoporosis (2, 3). The means by which resistance training achieves this is not fully understood. A study of paediatric patients with Inflammatory Bowel Disease found that this patient cohort tolerated high intensity exercise well (4). Regular exercise could help improve disease activity in Inflammatory Bowel Disease by the release of anti-inflammatory cytokines from myocytes during exercise.

Intestinal microbiota are now thought to be a key link in disease expression in humans (5). Previous studies have shown that aerobic exercise in obese adolescents has led to particular alterations in intestinal microbiota (6). These alterations appear to be related to the weight loss experienced. This may determine the quantity of weight and body fat lost by these adolescents.

Persistent resistance and aerobic exercise also leads to changes in baseline immunological profiles, particularly cytokines (7).

The investigators aim to explore the relationship between alterations in intestinal microbiota following a structured mixed cardio-respiratory and strength training exercise program and the correlation with changes on cytokine profile, percentage of body fat lost and disease activity.

Hypothesis:

1. A structured, 8-week mixed cardio-respiratory and resistance training exercise program results in specific changes in intestinal microbiota in inactive disease populations.
2. For inactive individuals, changes in intestinal microbiota following an 8-week exercise program are associated with changes in immunological profile.
3. Adjusting for the amount of exercise performed, greater decreases in percentage body fat are associated with the presence of particular intestinal microbiota changes after exercise.
4. Enhanced disease control, mood and anxiety states occur following an 8-week exercise program. This is associated with changes in the intestinal microbiota and immunological profiles.

Study design:

* Prospective, randomized control trial
* Interventional

Following identification of appropriate patients and subsequent recruitment both IBD and RA patients will equally be randomized into 2 groups in a 1:1 ratio.

The first group will enter an 8-week exercise program immediately and be measured at timepoint 0 - week 0 - and timepoint 1 - week 8. The second group will enter a delayed 8-week exercise program having first completed an 8-week period maintaining their usual levels of low physical activity. These patients will be measured at timepoint 0 , timepoint 1 and timepoint 2.

Sample Size:

The investigators will seek to recruit participants in the following groups

1. Inflammatory Bowel Disease, Ulcerative Colitis and Crohn's - 30 patients total
2. Rheumatoid Arthritis - 30 patients

Randomization process:

Subjects will be randomized into 8-week exercise or 16-week usual physical activity + exercise groups by their selection of appropriately marked envelopes containing the group number they are to be recruited to. Subjects will be recruited on a 1:1 basis to 8 week study: 16-week study respectively. Randomization will occur at the initial screening visit and will be witnessed by the subject and by 2 investigators.

Intervention:

A minimum standardized, mixed cardio-respiratory and resistance training exercise program will attempted to be adhered to. An individualized exercise program will be delivered with safety in mind. This program will be suitable for beginners and will be based around a basic "couch to 5km" exercise plan identical to that used in our previous research study, the ExMET study. In our experience participants enjoyed this program and progressed well, despite their baseline inactivity. Subjects are allowed to progress further than this program but only under supervision of the gym instructor or investigators. Free weights will not be included in the exercise program. For resistance exercises subjects will initially be required to perform 1 to 2 sets of 8 to 12 repetitions of 70% of their 1 Repetition max. This will be increased to 3 sets of 8 to 12 repetitions. An appropriate warm up will be encouraged to minimize injury. Gym instructors will be available on site throughout the exercise program for assistance if individuals have queries regarding their exercise program, recording of activities on FITLINXX or gym machinery.

* Type of exercise: Aerobic and resistance training - Options include walking/running on treadmill, stationary cycling, cross trainer, stepper machine for aerobic training. Resistance exercises will comprise 6-8 different machine based exercises focusing on core muscle strength as well as upper and lower body muscle groups e.g. chest press, leg extensions.
* Intensity: Moderate to vigorous intensity as per the Borg perceived exertion scale.
* Duration: 18 to 20 - minute aerobic sessions initially escalating weekly guided by standard couch to 5km protocols.
* Frequency: Three training sessions per week.
* Length: 8 weeks.

Methodology:

After recruitment, completion of the informed consent process and screening for inclusion and exclusion criteria, patients will be asked to attend 2 or 3 measurement visits depending on randomization. These visits will take place in the Clinical Sciences Building of Cork University Hospital. Confidential demographic data will be collected from each subject, including subject's sex, age, race, weight and height. Information regarding medical history and current medical status of the subject will be obtained. Validated questionnaires on medication adherence i.e. the Morisky adherence scale, physical activity and self-perceived stress: Beck Depression Inventory, Hospital Anxiety and Depression scale and State/trait Anxiety Inventory questionnaires as well as quality of life questionnaires including the SF-36 will be filled out.

Dual-Energy X-ray Absorptiometry scanning will be conducted to measure body composition including percentage body fat.

Patients will complete a detailed dietary survey the Food Frequency Questionnaire similar to that carried out in a recent study from our centre (8). Disease activity of patients will be assessed through clinical exam and history. Disease activity index scores, Harvey Bradshaw for Crohn's Disease, Powell-Tuck for Ulcerative Colitis and DAS-28-CRP for RA will be recorded.

Following these measurements and an appropriate warm up, individuals will undergo the Rockport one-mile walk test to establish a baseline level of fitness and estimated VO2 max. This sub-maximal fitness test entails participants walking one mile at a brisk pace without stopping. They are timed and at the end of the procedure the individual's heart rate is measured. An estimated VO2 max can be calculated based on previous validated studies (9). This test will be conducted under consistent and reliable environmental conditions at the indoor track at the Mardyke Arena.

Following theses procedures and measurements, subjects will be familiarized with the exercise program and equipment within the Mardyke arena. Subjects will attend a 90-minute induction session with a dedicated gym instructor from the Mardyke Arena. During these sessions the instructors will demonstrate the safe and appropriate use of equipment, illustrating the correct technique for resistance exercises. In order to keep a record of all exercise sessions conducted during the 8-week exercise programs, participants will be shown how to correctly record their individual activity on the FITLINXX activity monitoring system, adjacent to each machine in the Mardyke Arena. Subjects will have ample opportunity to try out and practice on these machines as well as being measured for their 1 repetition max. values required for the individual muscle strengthening goals.

Training program compliance will be monitored by examining weekly downloads of each subject's logged exercise activities in the Mardyke arena. For those subjects not maintaining the minimum exercise requirements, the subject will be contacted by telephone and facilitated to ensure progress matches the minimum standard over the following week. If this is not achieved or the subject wishes to withdraw from the study, they will no longer be involved in the study.

Outcome measures:

* Change in Intestinal Microbiota and virome - Intestinal microbiota and virome will be sampled from faecal samples provided by the subjects. These will then be stored before being characterized and quantified. Bile acid profiles (faecal, blood and urinary profiles) will be analyzed at beginning and end of study to see for potential changes with exercise. This will be performed in the APC, University College Cork or Teagasc Moorepark, Fermoy.
* Resting levels of immunological markers (cytokines such as TNF alpha, IL-6) at time points during the program.
* Change in glucose and cholesterol profiles in response to exercise.
* Proof of change in fitness - Predicted VO2 max via 1-mile walk test (Rockport test).
* Change in percentage body fat - DEXA - Total body composition scans performed in CUH.
* Basic Biochemistry and Haematology including CRP and creatine kinase
* Weight, height, BMI and waist/hip measurements.
* Food frequency diary including alcohol consumption to be measured at week 0 and week 8.
* Urinary, faecal and blood microbial metabolomics measured at each timepoint
* Disease activity scores - these will be measured by validated disease activity indices; Harvey-Bradshaw Index for patients with Crohn's Disease and the Simple Clinical Colitis Activity Index as well as the and Powell-Tuck Index for patients with Ulcerative Colitis. For patients with RA the DAS-28 CRP score will be calculated.
* Quality of life, mood and Anxiety Scores will be recorded: The Beck depression inventory, Hospital Anxiety and Depressions Scale (HADS), the State/Trait Anxiety Inventory will be used to monitor changes in mood/ anxiety. The Short form-36 (SF 36) will be used to monitor quality of life change.

Overall Statistical Data Analysis:

The investigators have access to sophisticated biostatistical analysis platforms for generating associations based upon diverse criteria.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 40 year-old male and females
* BMI between 22 and 35
* Confirmed diagnosis of Crohn's Disease, Ulcerative Colitis or Rheumatoid Arthritis
* Currently inactive i.e. No involvement in regular organized physical activity and with low weekly physical activity levels - as defined by the International Physical Activity Questionnaire (IPAQ)
* No regular organized physical activity in the last month
* Subject is willing to comply thoroughly with the basic, standard requirements of the training program
* Subject is willing to refrain from taking any unspecified dietary, probiotics, multivitamin or herbal supplements (14-day washout period pre-commencement of exercise program)
* Participant is happy to confine their formal exercise to within the Mardyke Arena
* Deemed to be fit to participate in exercise program for 8 weeks by the study investigators

Exclusion Criteria:

* History of coronary artery disease, congenital heart disease or any cardiovascular disease, including a family history of coronary artery disease before 45 years of age
* Uncontrolled hypertension (>140/90mmHg) (not white coat)
* Course of antibiotics or bowel preparation for endoscopy one month prior to the commencement of the exercise program
* Psychiatric disorders
* Any medical condition deemed exclusionary by the Principle Investigator
* A history of substance abuse
* History of total colectomy
* Currently treated with high dose corticosteroids or disease flare within 2 weeks of starting exercise program
* Pregnant
* History of faecal incontinence
* Have a malignant disease or any concomitant end stage organ disease
* Patients may not be receiving any experimental drug or have been involved in a recent experimental trial in the last 30 days

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Body composition alterations in patients with exercise. | 8 weeks
  To determine the metabolic and body composition alterations that occur in these patients with exercise as measured by changes in body fat composition measured using DEXA imaging and relate these changes to microbiota change

SECONDARY OUTCOMES:
Changes in fecal bile acids | 8 weeks
  Patinets fecal bile acids will be measured pre and post intervention
Changes in markers of intestinal inflammation (faecal calprotectin) that occur with exercise | 8 weeks
  Changes in markers of intestinal inflammation (faecal calprotectin) that occur with exercise will be measured
Alterations in gut microbiota | 8 weeks
  To compare alterations in gut microbiota following similar levels of exercise to previously recruited and exercised controls (The ExMET study)
Impact of medium-term moderate intensity exercise on resting inflammatory profiles (cytokines) in these patients. | 8 weeks
Changes in Harvey Bradshaw index in subjects with Crohn's disease | 8 weeks
  In subjects with Crohn's disease we will determine if exercise leads to changes in disease activity as determined by the Harvey Bradshaw disease activity score.
Changes in Powell tuck score in subjects with ulcerative colitis | 8 weeks
  In subjects with ulcerative colitis we will determine if exercise leads to changes in disease activity score as determined by the Powell tuck score
Changes in DAS-28 CRP score in subjects with rheumatoid arthritis | 8 weeks
  In subjects with rheumatoid arthritis we will determine if exercise leads to changes in disease activity scores as determined by the DAS-28 CRP score.
Changes in Predicted VO2 max via 1-mile walk test (Rockport test) | 8 weeks
  Changes in physical fitness as determined using predicted VO2 max via 1-mile walk test (Rockport test) resulting from the intervion will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Fergus Shanahan, MD, DSc., Principal Investigator — Professor and Chair Dept. of Medicine, University College Cork
Locations (1):
- Alimentary Pharmabiotic Centre, University College Cork, Cork, Cork, Ireland

REFERENCES:
- [Background] Hotamisligil GS. Inflammation and metabolic disorders. Nature. 2006 Dec 14;444(7121):860-7. doi: 10.1038/nature05485. PMID 17167474
- [Background] Zhao G, Li C, Ford ES, Fulton JE, Carlson SA, Okoro CA, Wen XJ, Balluz LS. Leisure-time aerobic physical activity, muscle-strengthening activity and mortality risks among US adults: the NHANES linked mortality study. Br J Sports Med. 2014 Feb;48(3):244-9. doi: 10.1136/bjsports-2013-092731. Epub 2013 Oct 4. PMID 24096895
- [Background] Siegrist M. [Role of physical activity in the prevention of osteoporosis]. Med Monatsschr Pharm. 2008 Jul;31(7):259-64. German. PMID 18808074
- [Background] Prakash S, Rodes L, Coussa-Charley M, Tomaro-Duchesneau C. Gut microbiota: next frontier in understanding human health and development of biotherapeutics. Biologics. 2011;5:71-86. doi: 10.2147/BTT.S19099. Epub 2011 Jul 11. PMID 21847343
- [Background] Santacruz A, Marcos A, Warnberg J, Marti A, Martin-Matillas M, Campoy C, Moreno LA, Veiga O, Redondo-Figuero C, Garagorri JM, Azcona C, Delgado M, Garcia-Fuentes M, Collado MC, Sanz Y; EVASYON Study Group. Interplay between weight loss and gut microbiota composition in overweight adolescents. Obesity (Silver Spring). 2009 Oct;17(10):1906-15. doi: 10.1038/oby.2009.112. Epub 2009 Apr 23. PMID 19390523
- [Background] de Salles BF, Simao R, Fleck SJ, Dias I, Kraemer-Aguiar LG, Bouskela E. Effects of resistance training on cytokines. Int J Sports Med. 2010 Jul;31(7):441-50. doi: 10.1055/s-0030-1251994. Epub 2010 Apr 29. PMID 20432196
- [Background] Claesson MJ, Jeffery IB, Conde S, Power SE, O'Connor EM, Cusack S, Harris HM, Coakley M, Lakshminarayanan B, O'Sullivan O, Fitzgerald GF, Deane J, O'Connor M, Harnedy N, O'Connor K, O'Mahony D, van Sinderen D, Wallace M, Brennan L, Stanton C, Marchesi JR, Fitzgerald AP, Shanahan F, Hill C, Ross RP, O'Toole PW. Gut microbiota composition correlates with diet and health in the elderly. Nature. 2012 Aug 9;488(7410):178-84. doi: 10.1038/nature11319. PMID 22797518
- [Background] Curatolo P, Giuffre R. [Dermal cranial sinuses in childhood and adolescence]. Minerva Pediatr. 1977 Dec 15;29(39):2357-61. No abstract available. Italian. PMID 600239
- [Background] Breen EC, Reynolds SM, Cox C, Jacobson LP, Magpantay L, Mulder CB, Dibben O, Margolick JB, Bream JH, Sambrano E, Martinez-Maza O, Sinclair E, Borrow P, Landay AL, Rinaldo CR, Norris PJ. Multisite comparison of high-sensitivity multiplex cytokine assays. Clin Vaccine Immunol. 2011 Aug;18(8):1229-42. doi: 10.1128/CVI.05032-11. Epub 2011 Jun 22. PMID 21697338
- [Derived] Cronin O, Barton W, Moran C, Sheehan D, Whiston R, Nugent H, McCarthy Y, Molloy CB, O'Sullivan O, Cotter PD, Molloy MG, Shanahan F. Moderate-intensity aerobic and resistance exercise is safe and favorably influences body composition in patients with quiescent Inflammatory Bowel Disease: a randomized controlled cross-over trial. BMC Gastroenterol. 2019 Feb 12;19(1):29. doi: 10.1186/s12876-019-0952-x. PMID 30755154